CLINICAL TRIAL: NCT02452164
Title: Family MobilePhone Otoscopy in Diagnostics of Otitis Media. (Family mOTO-Study)
Brief Title: Family MobilePhone Otoscopy in Diagnostics of Otitis Media
Acronym: FamilymOTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: T91/2015
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Otitis Media
Keywords: otoscopy; otitis media; cellphone; family
MeSH Terms: conditions — Otitis Media | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teaching group (Active Comparator): Parents are taught to conduct cellphone otoscopy and if necessary study physician removes cerumen from childrens´ ear canals at the first study visit.
  Interventions: Other: Teaching; Device: (CellScopeOTO)
- Control group (Other): Families receive the cellphone otoscope as if they had bought it themselves from the internet. After the first study week, parents are taught to conduct cellphone otoscopy and if necessary study physician removes cerumen from childrens´ ear canals.
  Interventions: Device: (CellScopeOTO)

INTERVENTIONS:
Other: Teaching
  Arms: Teaching group
Device: (CellScopeOTO)

SUMMARY:
This is a one-center clinical study carried out in Turku, Finland. The study patients will be randomly allocated to one of the two parallel study groups (teaching group and control group). The hypothesis is that the diagnostic quality of tympanic membrane imagines is better when parents have been taught to conduct middle ear examination with a cellphone otoscope (CellScopeOTO) as compared to no teaching. Furthermore, this study aims at evaluating the diagnostic feasibility of cellphone otoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 - 35 mo
* Parents have iPhone 5, 5s or 6
* Child is in daycare
* Child has had at least one acute otitis media within 90 days preceding the enrollment
* Family agrees to give a mortgage of 40 euros from the CellScopeOTO

Exclusion Criteria:

* Tympastonomy tube present in tympanic membrane
* Chronic perforation of the tympanic membrane
* Condition of head/neck anomaly to affect middle ear or ear canal anatomy
* One child from the family already participating

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
diagnostic quality of tympanic membrane imagines | first study week
  diagnostic quality of tympanic membrane imagines obtained by parents with cellphone otoscope

CONTACTS AND LOCATIONS:
Overall Officials: Aino Ruohola, MD, PhD, Principal Investigator — consultant
Locations (1):
- Turku University Hospital, Turku, Finland